CLINICAL TRIAL: NCT02607384
Title: A School-based Intervention to Diagnose and Treat Vision Problems in Elementary School Children With Reading Difficulty
Brief Title: The Baltimore Reading and Eye Disease Study
Acronym: BREDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00032063
Record Dates: First submitted 2015-11-12; First posted 2015-11-18 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Refractive Error; Visual Impairment; Convergence Insufficiency; Reading Disabilities
MeSH Terms: conditions — Refractive Errors; Vision Disorders; Ocular Motility Disorders; Dyslexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vision problems (Experimental): Children with refractive error will be prescribed eyeglass wearing, and children with convergence insufficiency will be given orthoptic exercises. Children with any other vision problem will be given a specialist referral to a pediatric eye specialist.
  Interventions: Behavioral: Eyeglass wearing; Behavioral: Orthoptic exercises; Other: Specialist referral

INTERVENTIONS:
Behavioral: Eyeglass wearing — Children found to require eyeglasses will be given two pairs free of charge
Behavioral: Orthoptic exercises — Children found to have convergence insufficiency will be prescribed orthoptic exercises
Other: Specialist referral — Children found to any other eye condition will be referred to a pediatric eye care specialist

SUMMARY:
The Baltimore Reading and Eye Disease Study (BREDS) is a two year study to determine the prevalence of vision problems in an early school age population with reading difficulty. Comprehensive vision and reading tests will be administered to 400 students at participating schools in the Baltimore City Public School system.

A secondary goal is to examine the impact of vision treatment on reading performance. Children with refractive error or convergence insufficiency will be provided treatment free of charge. The investigators will evaluate the impact that the treatment has on vision function and reading performance.

DETAILED DESCRIPTION:
Learning to read is a fundamental skill taught in the early years of elementary school education. Students who experience difficulty reading are at risk for long-term struggles with academic achievement. In fact, achieving reading proficiency by the end of third grade has been established as key predictor of life success.

While a number of factors contribute to reading problems, an undiagnosed or untreated ocular condition may present one possible etiology. To the investigator's knowledge, there are no large scale or prospective studies evaluating the prevalence of vision disorders in children with reading difficulties. Previously, the Baltimore Pediatric Eye Disease Study performed visual assessments in the Baltimore area for children 6 months through 5 years of age to establish the prevalence of select ocular disorders in this pre-school population. Little is known about the types of vision problems that affect a grade school population with and without reading difficulty.

There is general consensus that undiagnosed or untreated vision problems may contribute to reading difficulty, although the extent to which treatment will improve reading performance is not well established. Although there are some studies demonstrating that treatment of vision problems can improve reading performance, publications on the efficacy of school-based interventions to identify and treat vision problems in school-age children are lacking. If successful, a school-based intervention could have significant impact improving reading performance, especially in high poverty neighborhoods where children have the highest risk of poor reading aptitude and limited access to eye care services.

The primary goal of this research study is to determine the prevalence of vision problems in an early school age population with reading difficulty. To adequately address this question, the investigators will administer reading and vision assessments to 400 second and third graders in participating schools within the Baltimore City Public School system. In addition, the investigators will obtain information on how many children with vision problems have received treatment in the past, and if not, why not. The investigators will also determine how schools handle and refer children who are felt to be poor readers in order to assist with planning future interventions.

This study will be conducted over a two-year period. In the first year, the investigators conducted baseline vision and reading assessment on all participating subjects. In the second year, the investigators will conduct follow up vision and reading assessments on all children treated with eyeglasses or eye exercises and a subset of subjects with healthy eye exams. The investigators plan to evaluate any barriers to interventions, and where possible assist in overcoming such barriers, for example by replacing lost/broken eyeglasses.

A secondary goal is to examine the impact of vision treatment on reading performance. Children with refractive error and convergence insufficiency will be provided treatment free of charge. The investigators will evaluate the impact that the treatment has on vision function and reading performance.

In subsequent phases of this project, the investigators also hope to learn how novel treatments (e.g. iPads) impact reading performance.

ELIGIBILITY:
Inclusion Criteria:

* Medically and cognitively capable of completing a reading test and eye examination

Exclusion Criteria:

* Limited English proficiency (as categorized by the school district)
* Severe cognitive delay that limits ability to complete a written examination
* Ocular condition that has resulted in severe, irreversible visual impairment
* Medical/ neurological co-morbidities causing significant cognitive delay or cortical visual impairment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of refractive error and convergence insufficiency among students who perform poorly on reading tests as measured by the Woodcock-Johnson III Tests of Achievement and Gray Oral Reading Test 4 (GORT-4). | 1 year
Association between refractive error and convergence insufficiency and reading ability as measured by the Woodcock-Johnson III Tests of Achievement and Gray Oral Reading Test 4 (GORT-4). | 2 years
Effect of correction of refractive error and orthoptic exercises on reading ability as measured by the Woodcock-Johnson III Tests of Achievement and Gray Oral Reading Test 4 (GORT-4). | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David S Friedman, MD, MPH, PhD, Principal Investigator — Johns Hopkins University; Megan E Collins, MD, Principal Investigator — Johns Hopkins University

REFERENCES:
- [Background] Francis DJ, Shaywitz SE, Stuebing KK, Shaywitz BA, & Fletcher, J. M. Developmental lag versus deficit models of reading disability: A longitudinal, individual growth curves analysis. Journal of Educational Psychology 1996; 88:3-17.
- [Background] Handler SM, Fierson WM, Section on Ophthalmology; Council on Children with Disabilities; American Academy of Ophthalmology; American Association for Pediatric Ophthalmology and Strabismus; American Association of Certified Orthoptists. Learning disabilities, dyslexia, and vision. Pediatrics. 2011 Mar;127(3):e818-56. doi: 10.1542/peds.2010-3670. Epub 2011 Feb 28. PMID 21357342
- [Background] Giordano L, Friedman DS, Repka MX, Katz J, Ibironke J, Hawes P, Tielsch JM. Prevalence of refractive error among preschool children in an urban population: the Baltimore Pediatric Eye Disease Study. Ophthalmology. 2009 Apr;116(4):739-46, 746.e1-4. doi: 10.1016/j.ophtha.2008.12.030. Epub 2009 Feb 25. PMID 19243832
- [Background] Friedman DS, Repka MX, Katz J, Giordano L, Ibironke J, Hawes P, Burkom D, Tielsch JM. Prevalence of decreased visual acuity among preschool-aged children in an American urban population: the Baltimore Pediatric Eye Disease Study, methods, and results. Ophthalmology. 2008 Oct;115(10):1786-95, 1795.e1-4. doi: 10.1016/j.ophtha.2008.04.006. Epub 2008 Jun 5. PMID 18538407
- [Background] Williams WR, Latif AH, Hannington L, Watkins DR. Hyperopia and educational attainment in a primary school cohort. Arch Dis Child. 2005 Feb;90(2):150-3. doi: 10.1136/adc.2003.046755. PMID 15665167
- [Background] Stifter E, Burggasser G, Hirmann E, Thaler A, Radner W. Monocular and binocular reading performance in children with microstrabismic amblyopia. Br J Ophthalmol. 2005 Oct;89(10):1324-9. doi: 10.1136/bjo.2005.066688. PMID 16170125
- [Background] Butler BC, Klein R. Inattentional blindness for ignored words: comparison of explicit and implicit memory tasks. Conscious Cogn. 2009 Sep;18(3):811-9. doi: 10.1016/j.concog.2009.02.009. Epub 2009 Mar 26. PMID 19328012
- [Background] Granet DB. Learning disabilities, dyslexia, and vision: The role of the pediatric ophthalmologist. J AAPOS. 2011 Apr;15(2):119-20. doi: 10.1016/j.jaapos.2011.03.003. No abstract available. PMID 21596289
- [Background] Levine MD. Reading disability: do the eyes have it? Pediatrics. 1984 Jun;73(6):869-70. No abstract available. PMID 6728588
- [Background] Lubkin V. The ophthalmologist and the reading problem. Bull N Y Acad Med. 1968 Apr;44(4):459-69. No abstract available. PMID 5241254
- [Background] Dusek WA, Pierscionek BK, McClelland JF. An evaluation of clinical treatment of convergence insufficiency for children with reading difficulties. BMC Ophthalmol. 2011 Aug 11;11:21. doi: 10.1186/1471-2415-11-21. PMID 21835034
- [Background] Borsting E, Mitchell GL, Kulp MT, Scheiman M, Amster DM, Cotter S, Coulter RA, Fecho G, Gallaway MF, Granet D, Hertle R, Rodena J, Yamada T; CITT Study Group. Improvement in academic behaviors after successful treatment of convergence insufficiency. Optom Vis Sci. 2012 Jan;89(1):12-8. doi: 10.1097/OPX.0b013e318238ffc3. PMID 22080400
- [Background] Heckman JJ. The case for investing in disadvantaged young children. Investing in our nation's future. First Focus Report 2008; 49-59
- [Derived] Huang AH, Guo X, Mudie LI, Wolf R, Owoeye J, Repka MX, Friedman DS, Slavin RE, Collins ME. Baltimore Reading and Eye Disease Study (BREDS): compliance and satisfaction with glasses usage. J AAPOS. 2019 Aug;23(4):207.e1-207.e6. doi: 10.1016/j.jaapos.2019.01.018. Epub 2019 May 18. PMID 31112777